CLINICAL TRIAL: NCT01082731
Title: A Multi-center, Open-label, Randomized, Phase 4, Trial of Artemether-Lumefantrine and Mefloquine-Artesunate for the Treatment of Uncomplicated P. Falciparum Malaria Parasitemia in Pregnant Women in Brazil
Brief Title: Efficacy of Artemisinin Combination Therapies for the Treatment of Uncomplicated P. Falciparum in Pregnancy in Brazil
Acronym: PAACT-PF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Extremely slow enrollment
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAACT-PF
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium falciparum; Treatment; Brazil
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mefloquine- Artesunate (Experimental): Mefloquine- Artesunate (Farmaguinhos, Brazil): tablets of 100 mg artesunate and 220 mg mefloquine (fixed dose combination), given once daily for 3 days.
  Interventions: Drug: Mefloquine- Artesunate
- Artemether- Lumefantrine (Active Comparator): Artemether-Lumefantrine: 4 tablets containing 20 mg of artemether plus 120 mg of lumefantrine per tablet twice daily for three days as 2 doses 8 hours apart on the 1st day and then 2 doses 12 hours apart on the 2nd and 3rd days, administered with a fatty meal
  Interventions: Drug: Artemether-Lumefantrine

INTERVENTIONS:
Drug: Artemether-Lumefantrine — 4 tablets containing 20 mg of artemether plus 120 mg of lumefantrine per tablet twice daily for three days as 2 doses 8 hours apart on the 1st day and then 2 doses 12 hours apart on the 2nd and 3rd days, administered with a fatty meal
  Other Names: Coartem; Lumet
  Arms: Artemether- Lumefantrine
Drug: Mefloquine- Artesunate — Tablets of 100 mg artesunate and 220 mg mefloquine (fixed dose combination), given once daily for 3 days.
  Other Names: Mefloquine- Artesunate (Farmaguinhos, Brazil)
  Arms: Mefloquine- Artesunate

SUMMARY:
Data on the burden of MIP in low transmission areas, such as Latin America, are very limited; there is even less information on the efficacy of case management of MiP. The treatment recommendations for MiP in Latin American countries have been changing rapidly in recent months; currently, either artemether-lumefantrine (AL) or mefloquine-artesunate (MA) is the first line treatment for P. falciparum (depending on country); however, no data exists on the efficacy of these drugs for the treatment of malaria in pregnancy in Latin America to support their use.

We propose a multi-center 2-arm open-label randomized Phase 4 clinical trial to assess safety and efficacy of the present therapies, AL and MA. We hypothesize that the drugs will both be efficacious for use in pregnant women in Brazil.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age >16 weeks (determined by LMP and fundal height)- if there is discordance between the two, the more conservative estimate (i.e. lower) will be used, to prevent accidental exposure of a 1st trimester fetus
2. Normal fetal heart beat detected by Doppler
3. Presence of any P. falciparum parasitemia ≤ 50,000 parasites/microliter (thick film)
4. Willing to sign or thumb print informed consent
5. Willing to return for scheduled follow up visits for treatment and observation until delivery
6. Willing to deliver in health facility

Exclusion Criteria:

1. Pregnancy < 16 weeks
2. Microscopically confirmed P. vivax or mixed infection/ parasitemia (P. falciparum and another species of Plasmodium, i.e. P. vivax, P. ovale, or P. malariae)
3. History of allergy or hypersensitivity to interventional drugs
4. Exposure to antimalarial drugs and other drugs with antimalarial activity within the past 2 months, as determined by history from the woman (quinine, mefloquine, or artemisinin derivatives, including AL and MA)
5. Patients taking drugs with possible interaction with study drugs (ie. warfarin, digoxin)
6. History or family history of epilepsy or psychiatric disorder
7. Presence of signs and symptoms of severe malaria
8. Hemoglobin < 7 g/dl
9. Inability to tolerate oral medication (repeated vomiting, impairment of consciousness).
10. History of chronic disease including diabetes, renal failure, hepatic failure, heart disease requiring anti-arrhythmic drugs or warfarin, HIV or AIDS, known hemoglobinopathy
11. Participant's inability to return for follow up visits
12. Age <15 years

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
63-day PCR-adjusted parasitological cure of P. falciparum | 63 days

CONTACTS AND LOCATIONS:
Overall Officials: Meghna Desai, PhD MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- Brazil (2):
  - Hospital Geral Maternidade de Cruzeiro do Sul, Cruzeiro do Sul, Acre
  - Centro de Pesquisa em Patologias Tropicais, Porto Velho, Rondônia